CLINICAL TRIAL: NCT05099133
Title: A Phase 1, Single-center, Double-blind, Randomized, Placebo-controlled, Single Ascending Dose Trial to Evaluate Pharmacokinetics, Immunogenicity, Safety, and Tolerability of LEO 138559 in Healthy Japanese Subjects
Brief Title: A Trial to Evaluate Pharmacokinetics, Immunogenicity, Safety, and Tolerability of LEO 138559 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0145-1486
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2022-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LEO 138559 Dose 1 (Experimental): LEO 138559 will be administered subcutaneously up to 3 injections per dosing
  Interventions: Drug: LEO 138559
- LEO 138559 Dose 2 (Experimental): LEO 138559 will be administered subcutaneously up to 3 injections per dosing
  Interventions: Drug: LEO 138559
- LEO 138559 Dose 3 (Experimental): LEO 138559 will be administered subcutaneously up to 3 injections per dosing
  Interventions: Drug: LEO 138559
- Placebo (Placebo Comparator): LEO 138559 placebo will be administered subcutaneously up to 3 injections per dosing
  Interventions: Drug: LEO 138559 Placebo

INTERVENTIONS:
Drug: LEO 138559 — LEO 138559 is an antibody given by injection just under the skin.
  Arms: LEO 138559 Dose 1; LEO 138559 Dose 2; LEO 138559 Dose 3
Drug: LEO 138559 Placebo — LEO 138559 placebo is given by injection just under the skin. LEO 138559 placebo contains the same excipients in the same concentration as LEO 138559, except the medical ingredient LEO 138559.
  Arms: Placebo

SUMMARY:
This trial will investigate the pharmacokinetics, immunogenicity, safety, and tolerability of LEO 138559 in healthy Japanese subjects.

The trial consists of a screening period of up to 4 weeks, a single treatment with either LEO 138559 or placebo, and 8 follow-up visits to Day 85.

A total of 24 healthy subjects will be enrolled in 3 dose groups (n=8 per dose group) and randomized to either LEO 138559 or placebo in a ratio of 6:2.

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 to 65 years of age, inclusive, at the Screening visit
2. Japanese subjects to be considered ethnic Japanese must:

   1. Be born in Japan with parents and grandparents (maternal and paternal) of Japanese descent
   2. Not have lived outside of Japan for more than 10 years at the time of Screening
   3. No significant change in lifestyle since leaving Japan, including diet.
3. Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive, at the Screening visit.
4. Healthy, determined by pre-trial medical evaluation at Principal Investigator's discretion

Exclusion Criteria

1. Female subjects of childbearing potential who are not willing to use highly effective contraception.
2. Subject has clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, immunological, musculoskeletal, infectious, metabolic, hematologic, neurological, or psychiatric disorder(s) as determined by the Principal Investigator or designee.
3. Subject has any surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of any drug as determined by the Principal Investigator or designee.
4. Clinically significant infection within 4 weeks prior to randomization that may compromise the safety of the subject in the trial or the integrity of the trial. This includes clinically significant infections (common cold is allowed [with negative SARS-CoV-2 PCR test]) that in the opinion of the Investigator or Sponsor's Medical Monitor may compromise the safety of the subject in the trial, interfere with evaluation of the IMP, or reduce the subject's ability to participate in the trial.
5. History of any active skin infection within 1 week prior to Screening or randomization.
6. Subject who has taken immunosuppressive/immunomodulating medication within 4 weeks prior to randomization, topical corticosteroids, topical calcineurin inhibitors within 2 weeks prior to randomization, or was treated with biologics within 5 half-lives (if known) or 12 weeks prior to randomization, whichever is longer.
7. Subject has used over-the-counter (OTC) medications (including vitamins), or herbal remedies from 14 days prior to admission until the End-of-trial Visit. By exception, paracetamol/acetaminophen ≤ 2 g per day is permitted.
8. History of chronic alcohol or drug abuse within 12 months prior to Screening, or any condition associated with poor compliance as judged by the Investigator.
9. Heavy smoker (daily average >10 cigarettes) within the last three months prior to Screening.
10. Subject is unwilling to avoid use of alcohol or alcohol-containing foods, medications, or beverages, within 36 hours prior to admission until discharge from the Clinical Unit.
11. Female subjects are breastfeeding or female subjects with a positive serum pregnancy test at the Screening visit or urine pregnancy test at admission.
12. Subject is unwilling to avoid consumption of coffee and caffeine-containing beverages within 48 hours prior to admission until discharge from the Clinical Unit.
13. Subject is unable to abstain from smoking (or other nicotine use) from admission until discharge from the Clinical Unit.
14. Subject scheduled to receive COVID-19 vaccination within 2 weeks before IMP administration.
15. Less than 4 weeks after the second COVID-19 vaccination or booster (if on a single dose vaccination, it should be 4 weeks after).
16. Live attenuated viral vaccine administration within 12 weeks before LEO 138559 or planned within three months after the last administration of LEO 138559.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
AUC0-last: the area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration | From Day 1 to Day 85
  Pharmacokinetic endpoint to be determined from serum concentrations
AUC0-inf: area under the concentration-time curve from pre-dose (time 0) extrapolated to infinite time | From Day 1 to Day 85
  Pharmacokinetic endpoint to be determined from serum concentrations
Cmax: maximum serum LEO 138559 concentration | From Day 1 to Day 85
  Pharmacokinetic endpoint to be determined from serum concentrations
tmax: time of maximum serum LEO 138559 concentration | From Day 1 to Day 85
  Pharmacokinetic endpoint to be determined from serum concentrations
t½: terminal elimination half-life | From Day 1 to Day 85
  Pharmacokinetic endpoint to be determined from serum concentrations
CL/F: apparent total body clearance | From Day 1 to Day 85
  Pharmacokinetic endpoint to be determined from serum concentrations
Vz/F: apparent volume of distribution | From Day 1 to Day 85
  Pharmacokinetic endpoint to be determined from serum concentrations

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | From Day 1 to Day 85
Presence of binding anti-drug antibodies | Day 1(pre-dose), Day 29, Day 57, and Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Investigational Site, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No